CLINICAL TRIAL: NCT01039012
Title: Tai Chi for Osteopenic Women: A Pilot Randomized Controlled Trial
Brief Title: Tai Chi for Osteopenic Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Harvard University Faculty of Medicine (Other)
Responsible Party: Peter M. Wayne, PhD, Assistant Professor of Medicine, Harvard Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT003503 (NIH)
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Osteopenia
Keywords: bone mineral density; osteoporosis; exercise; bone remodeling; biomotion analysis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Motor Activity | interventions — Tai Ji; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi plus Standard Care (Other)
  Interventions: Other: Tai Chi
- Standard Care (Other)
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Tai Chi — Participants randomized to the Tai Chi group select a Tai Chi school from a pre-screened list of community-based Tai Chi programs and enroll for 9 months. Participants are asked to attend classes twice a week for the first month and once a week for the remaining 8 months. They are also asked to practice at home, or attend more classes for 2-3 additional hours per week. While in the study they are also encouraged to follow the standard care as recommended by their physician.
  Arms: Tai Chi plus Standard Care
Other: Standard Care — Participant follow the standard care recommended by their physician.
  Arms: Standard Care

SUMMARY:
This study will assess the effectiveness of Tai Chi to affect the rate of bone loss in post-menopausal women who have been diagnosed with the initial stages of bone thinning.

DETAILED DESCRIPTION:
Osteopenia is a serious and growing public health concern for women. Osteopenic women are at greater risk for fractures than women with normal bone mineral densities (BMD). Low BMD-related fractures are associated with significant long-term impairment, high morbidity rates and high medical costs. Optimal preventive and sustainable interventions for osteopenic women are not yet well-defined.

Tai Chi, a mind-body exercise that is growing in popularity in the U.S., shows may be an effective, safe and practical intervention for women with low bone density. Preliminary studies suggest Tai Chi can reduce rates of BMD decline in post-menopausal women. While suggestive, these studies have numerous design limitations.

We propose a pilot randomized controlled trial to assess the efficacy and feasibility of Tai Chi as an adjunct to standard care for post-menopausal osteopenic women. Eight-six osteopenic women ages 45-70 will be recruited from a large multi-specialty group practice. Our primary aim is to assess the feasibility for recruiting and retaining osteopenic women into a randomized controlled trial of 9 months of Tai Chi. Our secondary aim is to collect preliminary data on the efficacy of Tai Chi in reducing rates of bone loss in osteopenic women using sensitive markers of bone turnover and dual-energy x-ray absorptiometry. The results of this study will inform the design of a future trial evaluating the benefits and safety for Tai Chi for osteopenic women, as well as the physiological and biomechanical mechanisms through which Tai Chi may impact BMD and fracture risks associated with osteopenia.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 45-70 years
* BMD T-scores of the hip (femoral neck or trochanter) and/or spine between -1.0 and -2.5
* Post-menopausal w/out menses for ≥ 12 months
* Sedentary, i.e. do not regularly participate in physical exercise on average 1 or more times per week

Exclusion Criteria:

* Osteoporotic (T-score < -2.5) or a fracture in the past 2 years not caused by motor vehicle accident
* Prior or current use of use of medication that increase risks of fracture (e.g. steroids, anti-convulsants, anticoagulants, lithium)
* Prior or current use of medications that modify bone metabolism (e.g. bisphosphonates, selective estrogen receptor modulators such as Raloxifene)
* Use of calcium supplements above levels suggested within the recommendations of standard care (i.e., above 1200-1500 mg)
* Current or prior year use of estrogen or calcitonin
* Malignancies other than skin cancer
* Diagnosis of anorexia along with a BMI of < 17.5
* Conditions that cause secondary osteoporosis (e.g. Cushing's syndrome, Marfan's syndrome)
* Tobacco use in past year
* Physical or mental disabilities that will preclude informed consent or active study participation
* Geographic or scheduling limitations that would preclude required participation in weekly Tai Chi classes and study procedures
* Current regular practice of Tai Chi

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Serum markers of bone resorption (CTX, C-terminal cross linking telopeptide of type I collagen), and bone formation (osteocalcin). | Baseline, 3 months, 9 months
Bone mass density of the lumbar spine and proximal femur (dual-energy X-ray absorptiometry). | Baseline, 9 months

SECONDARY OUTCOMES:
Secondary outcomes include health-related quality-of-life, exercise behavior, and psychological well-being. In addition, kinetic and kinematic characterization of gait, standing, and rising from a chair are assessed in subset of participants (n=16). | Baseline, 3 months, 9 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Wayne PM, Kiel DP, Buring JE, Connors EM, Bonato P, Yeh GY, Cohen CJ, Mancinelli C, Davis RB. Impact of Tai Chi exercise on multiple fracture-related risk factors in post-menopausal osteopenic women: a pilot pragmatic, randomized trial. BMC Complement Altern Med. 2012 Jan 30;12:7. doi: 10.1186/1472-6882-12-7. PMID 22289280
- [Derived] Wayne PM, Buring JE, Davis RB, Connors EM, Bonato P, Patritti B, Fischer M, Yeh GY, Cohen CJ, Carroll D, Kiel DP. Tai Chi for osteopenic women: design and rationale of a pragmatic randomized controlled trial. BMC Musculoskelet Disord. 2010 Mar 1;11:40. doi: 10.1186/1471-2474-11-40. PMID 20193083